CLINICAL TRIAL: NCT06388434
Title: Influence of Attentional Control on Protective Arm Responses to Balance Perturbations in Older Adults and People with Peripheral Neuropathy
Brief Title: Protective Arm Balance Responses
Acronym: PAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kelly Westlake, PI, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HP-00100309
Record Dates: First submitted 2023-07-11; First posted 2024-04-29 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Old Age; Debility; Peripheral Neuropathy
Keywords: Reactive Balance; Reach to Grasp; Attention Switching
MeSH Terms: conditions — Frailty; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The study will include two groups (older adults and people with peripheral neuropathy) which will be assessed pre- and post-intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Protective Arm Training (Experimental): Both groups (older adults and people with peripheral neuropathy) will be assessed pre- and post-intervention as well as midway through the training.
  Interventions: Behavioral: Protective Arm Balance Response Training

INTERVENTIONS:
Behavioral: Protective Arm Balance Response Training — Participants will be trained in the reach to grasp arm balance response while being exposed to unpredictable balance perturbations

SUMMARY:
The overall objective of this study is to investigate the effect of attention control training on reach-grasp stabilizing responses during fall-induced perturbations. The central hypothesis is that training attention control during reach to grasp balance perturbations will lead to increased grasp accuracies and reduced in-task falls. This research will mark the first explore the effects of training attention control on protective arm responses and fall rate during a balance perturbation paradigm and the first feasibility testing of a fully integrated cognitive and physical rehabilitation paradigm, moving beyond correlative designs and parallel treatments. The overall public health significance of the proposed research is that with improved protective arm responses and grasp accuracies, a larger randomized control study may be designed to mitigate falls among community dwelling older adults.

Participants will be involved in 6 sessions. Session 1 will include the assessment, questionnaires, and training. Session 2 will include just the training. Session 3 will include the assessment and training. Sessions 4-5 will include just the training. Session 6 will include the assessment, questionnaires, and training.

DETAILED DESCRIPTION:
Participants will be involved in 6 sessions. Session 1 will include the assessment, questionnaires, and training. Session 2 will include just the training. Session 3 will include the assessment and training. Sessions 4-5 will include just the training. Session 6 will include the assessment, questionnaires, and training.

Assessment:

Using a specialized treadmill that induces balance perturbations (ActiveStep, www.simbex.com), an individualized perceived balance threshold will first be assessed. In brief, participants will stand feet together, arms relaxed at their sides, eyes focused on a red 'X' at eye level and asked only to grasp when participants feel a true need to restore balance. Testing perturbations will proceed 2 levels above this threshold. Next, two lateral perturbation conditions, each with 10 trials (5x right; 5x left) will be randomly applied. Perturbation direction and timing will be unknown and random. Condition 1 has no cognitive task. Condition 2 has participants engaged in a cognitive task 30-120s prior to perturbation with instructions, "as soon as the participant feels a falling sensation, stop the task and grab a single rail to quickly restore balance." To promote high cognitive task engagement, a mental arithmetic task was selected as one of the most effective stressors. Psychophysiological stressors are known to result in greater task engagement than pleasant tasks, thus adding a consistent challenge to task inhibition and in turn, attention switching. To allow characterization of the 'first trial response', the first and second trial will include one of each condition, separated by a 5min rest. The 'first trial response' has less stability compared with subsequent perturbations and is relevant to the study of mechanisms underlying 'real-life' falls. Objective kinematic and electromyographic (EMG) assessment of balance responses to the perturbations will be conducted. Following the balance perturbation assessment, clinical tests of balance, including the four square step test and miniBEST, will be conducted. The investigators will also be using a device to record physiological responses using sensors attached to the fingers (Biopac Systems, Inc.) to record stress at baseline and during the reactive balance responses assessment.

Subjects will also complete questionnaires on balance confidence and anxiety. These include:

1. Activity specific balance confidence scale (ABC): Questions are on how confidence subjects feel when performing normal activities of daily living that involves maintaining their dynamic balance.
2. Stait Trait Anxiety Inventory: Measure of trait and state anxiety
3. Subjective Units of Distress Scale (SUDS): Measures anxiety and distress on a scale of 0 no distress and totally relaxed to 100 highest distress/ anxiety ever felt
4. Mini Mental State Examination (MMSE): A validated sensitive test for detecting mild cognitive impairments. It involves documenting the participants responses to cognitive tasks such as c subtractions, memory recall repeating number sequences, naming as many nouns starting with "F" etc.
5. Beck Anxiety Inventory (BAI): Consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week

Training:

Participants will each undergo 6 sessions of an attention task combined with balance perturbation and upper limb responses. The investigators define feasibility in terms of whether key components of our approach are met, including valid and reliable pre-perturbation cognitive engagement and reactive arm recovery responses over repeated trials, as well as overall participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 65 to 88 years of age
* Community ambulatory with or without a straight cane

Exclusion Criteria:

* Significant musculoskeletal or neurological impairments as indicated by limitations in activities of daily living, ADL (less than 6/6 on Katz Index in ADLs)
* Clinically identified uncorrected visual loss
* Complaints of dizziness or known vestibular disorder
* Upper extremity strength less than 4/5 manual muscle test at the shoulder, elbow, wrist, or grip.
* Mini Mental State Examination score of less than 25

Ages: 45 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Grasp Accuracy | Within the first second immediately following the balance perturbation onset
  Grasp accuracy refers to the success of the reach to grasp response. This can be a full grasp (grasping with all 5 fingers), overshoot, or undershoot of the handrail
In-task falls incidence | The peak load on the safety harness within the first second of the balance perturbation onset.
  A load cell attached to the overhead safety harness will record the percentage of the participants body weight that is being supported by the harness. If the harness is holding up more than 30% of the participants body weight, this is considered a fall, 4.5-30% of the participants body weight is considered a harness-assist, and less than 4.5% of the participants body weight is considered recovery.

SECONDARY OUTCOMES:
Electromyography (EMG) of the shoulder muscles | Within the first second following onset of the balance perturbation
  EMG will allow us to record muscle activity during the balance response
Physiological responses (heart rate variability) | 5 minutes at baseline and 5 minutes during the balance perturbation tasks
  Heart rate variability informs us about the ability of the heart to adapt to different stressors by calculating the variability in heart rate during different tasks.
Physiological responses (electrodermal activity) | 5 minutes at baseline and 5 minutes during the balance perturbation tasks
  Electrodermal activity informs us about the amount of stress in the body during various tasks by calculating the amount of sweat produced during the task (the more we sweat, the more stressed we are).
Activity specific balance confidence scale | The questions ask about the 4 weeks before the first day of testing
  Questions are on how confidence subjects feel when performing normal activities of daily living that involves maintaining their dynamic balance.
Stait Trait Anxiety Inventory | The questions ask about the participants current feelings and their feelings in general over the past year
  Measure of trait and state anxiety
Subjective Units of Distress Scale | In the moment immediately following the balance perturbations
  Measures anxiety and distress on a scale of 0 no distress and totally relaxed to 100 highest distress/ anxiety ever felt
Mini Mental State Examination (MMSE) | At baseline
  A validated sensitive test for detecting mild cognitive impairments. It involves documenting your responses to cognitive tasks such as subtractions, memory recall repeating number sequences, naming as many nouns starting with "F" etc.
Beck Anxiety Inventory | The items in the scale ask about the participants feelings over the previous week
  Consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week
Somatosensation | This will be assessed at baseline only
  Consists of a comprehensive assessment of somatosensation including proprioception, vibration, light touch, and protective sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly P Westlake, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Allied Health Research Building, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available if requested
Supporting Information: Study Protocol, SAP
Time Frame: Will be made available upon publication of results
Access Criteria: Access will be granted through the published article or upon reasonable request

REFERENCES:
- [Background] Stevens JA, Mahoney JE, Ehrenreich H. Circumstances and outcomes of falls among high risk community-dwelling older adults. Inj Epidemiol. 2014 Mar 20;1(5):5. doi: 10.1186/2197-1714-1-5. PMID 26744637
- [Background] Kim KJ, Ashton-Miller JA. Biomechanics of fall arrest using the upper extremity: age differences. Clin Biomech (Bristol). 2003 May;18(4):311-8. doi: 10.1016/s0268-0033(03)00005-6. PMID 12689781
- [Background] Marigold DS, Bethune AJ, Patla AE. Role of the unperturbed limb and arms in the reactive recovery response to an unexpected slip during locomotion. J Neurophysiol. 2003 Apr;89(4):1727-37. doi: 10.1152/jn.00683.2002. Epub 2002 Dec 11. PMID 12611998
- [Background] Hsiao ET, Robinovitch SN. Common protective movements govern unexpected falls from standing height. J Biomech. 1998 Jan;31(1):1-9. doi: 10.1016/s0021-9290(97)00114-0. PMID 9596532
- [Background] Hendriks MR, Bleijlevens MH, van Haastregt JC, Crebolder HF, Diederiks JP, Evers SM, Mulder WJ, Kempen GI, van Rossum E, Ruijgrok JM, Stalenhoef PA, van Eijk JT. Lack of effectiveness of a multidisciplinary fall-prevention program in elderly people at risk: a randomized, controlled trial. J Am Geriatr Soc. 2008 Aug;56(8):1390-7. doi: 10.1111/j.1532-5415.2008.01803.x. Epub 2008 Jul 24. PMID 18662214
- [Background] Province MA, Hadley EC, Hornbrook MC, Lipsitz LA, Miller JP, Mulrow CD, Ory MG, Sattin RW, Tinetti ME, Wolf SL. The effects of exercise on falls in elderly patients. A preplanned meta-analysis of the FICSIT Trials. Frailty and Injuries: Cooperative Studies of Intervention Techniques. JAMA. 1995 May 3;273(17):1341-7. PMID 7715058
- [Background] Mansfield A, Wong JS, Bryce J, Knorr S, Patterson KK. Does perturbation-based balance training prevent falls? Systematic review and meta-analysis of preliminary randomized controlled trials. Phys Ther. 2015 May;95(5):700-9. doi: 10.2522/ptj.20140090. Epub 2014 Dec 18. PMID 25524873
- [Background] Bolton DAE, Patel R, Staines WR, McIlroy WE. Transient inhibition of primary motor cortex suppresses hand muscle responses during a reactive reach to grasp. Neurosci Lett. 2011 Oct 24;504(2):83-87. doi: 10.1016/j.neulet.2011.09.001. Epub 2011 Sep 10. PMID 21925570
- [Background] Liston C, McEwen BS, Casey BJ. Psychosocial stress reversibly disrupts prefrontal processing and attentional control. Proc Natl Acad Sci U S A. 2009 Jan 20;106(3):912-7. doi: 10.1073/pnas.0807041106. Epub 2009 Jan 12. PMID 19139412
- [Background] Sanger J, Bechtold L, Schoofs D, Blaszkewicz M, Wascher E. The influence of acute stress on attention mechanisms and its electrophysiological correlates. Front Behav Neurosci. 2014 Oct 9;8:353. doi: 10.3389/fnbeh.2014.00353. eCollection 2014. PMID 25346669
- [Background] Cheng KC, Pratt J, Maki BE. Effects of spatial-memory decay and dual-task interference on perturbation-evoked reach-to-grasp reactions in the absence of online visual feedback. Hum Mov Sci. 2013 Apr;32(2):328-42. doi: 10.1016/j.humov.2012.11.001. Epub 2013 Apr 29. PMID 23635599
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Padgett PK, Jacobs JV, Kasser SL. Is the BESTest at its best? A suggested brief version based on interrater reliability, validity, internal consistency, and theoretical construct. Phys Ther. 2012 Sep;92(9):1197-207. doi: 10.2522/ptj.20120056. Epub 2012 Jun 7. PMID 22677295
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Daniels JK, McFarlane AC, Bluhm RL, Moores KA, Clark CR, Shaw ME, Williamson PC, Densmore M, Lanius RA. Switching between executive and default mode networks in posttraumatic stress disorder: alterations in functional connectivity. J Psychiatry Neurosci. 2010 Jul;35(4):258-66. doi: 10.1503/jpn.090175. PMID 20569651
- [Background] Kim HG, Cheon EJ, Bai DS, Lee YH, Koo BH. Stress and Heart Rate Variability: A Meta-Analysis and Review of the Literature. Psychiatry Investig. 2018 Mar;15(3):235-245. doi: 10.30773/pi.2017.08.17. Epub 2018 Feb 28. PMID 29486547
- [Background] Andersson S, Finset A. Heart rate and skin conductance reactivity to brief psychological stress in brain-injured patients. J Psychosom Res. 1998 Jun;44(6):645-56. doi: 10.1016/s0022-3999(97)00305-x. PMID 9678746
- [Background] Carriere JSA, Seli P, Smilek D. Wandering in both mind and body: individual differences in mind wandering and inattention predict fidgeting. Can J Exp Psychol. 2013 Mar;67(1):19-31. doi: 10.1037/a0031438. PMID 23458548